CLINICAL TRIAL: NCT07022496
Title: Assessment of Oral Caffeine Intake in Reducing the Severity of Acute Migraine Attack Among Patients Attending Headache and Neurology Outpatients Clinic of Ainshams University Hospitals: A Randomized Controlled Trial
Brief Title: Assessment of Oral Caffeine Intake in Changing the Severity of Acute Migraine Attack Using VAS Score Among Patients Attending Headache and Neurology Outpatients Clinic of Ainshams University Hospitals
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nourhan Nader, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD87/2023
Record Dates: First submitted 2024-12-23; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Migraine Disease; Migraine Headache; Migraine Headache, With or Without Aura; Migraine, Acute
MeSH Terms: conditions — Migraine Disorders | interventions — Caffeine; Tryptamines; Anti-Inflammatory Agents, Non-Steroidal; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine group (Experimental): Caffeine group added to standard treatment
  Interventions: Drug: Caffeine (200 mg); Drug: triptans; Drug: NSAID (Nonsteroidal anti-inflammatory drugs); Drug: Paracetamol (acetaminophen)
- Control group (Active Comparator): Standard treatment (NSAIDS, Triptans, or Acetaminophen)
  Interventions: Drug: triptans; Drug: NSAID (Nonsteroidal anti-inflammatory drugs); Drug: Paracetamol (acetaminophen)

INTERVENTIONS:
Drug: Caffeine (200 mg) — caffeine tablets
  Arms: Caffeine group
Drug: triptans — Sumatriptan
Drug: NSAID (Nonsteroidal anti-inflammatory drugs) — Aspirin 250 mg, 81 mg, 75 mg
Drug: Paracetamol (acetaminophen) — Paracetamol 250 mg

SUMMARY:
Caffeine extracted from green tea to abort acute attack of Migraine

DETAILED DESCRIPTION:
Caffeine tablets extracted from green tea can be used as caffeinated drinks to decrease intensity of migraine attacks

ELIGIBILITY:
Inclusion Criteria:

Patients suffering from migraine with aura, migraine without aura, episodic, and chronic migraine according to ICHD-3 diagnosis will be legible for the study.

Exclusion Criteria:

Patients who have history of any cardiac dysrhythmia, hypertension, ischemic heart disease, active peptic ulcer disease, inflammatory bowel disease, obsessive compulsive disorder, pregnancy, breast-feeding, renal failure, hepatic failure, sleep disorder, mental retardation, and history of substance abuse that prevent them from cooperating with us during the study Patients who had headache due to: Cluster headache, trigeminal neuralgia, glossopharyngeal neuralgia, headache secondary to trauma, cranial disorder, vascular disorder, infection, or mass lesion, will also be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To reduce the severity of migraine attack | Three years
  using Visual analogue scale

SECONDARY OUTCOMES:
To evaluate the effect of oral caffeine in reducing pain associated with acute migraine attacks among patients attending Headache Clinic, Ain Shams University hospital via Visual analogue scale | Three year
  To assess the pain reduction through visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Abstract